CLINICAL TRIAL: NCT01297660
Title: Neuro-urological Outcome After Spinal Cord Injury
Status: Completed | Type: Observational
Sponsor: Balgrist University Hospital (Other)
Responsible Party: Principal Investigator, Thomas Kessler, PD Dr. med., Balgrist University Hospital
Other Study IDs: KEK-2010-0207/01
Record Dates: First submitted 2011-02-16; First posted 2011-02-17 (Estimated); Last update posted 2016-12-16 (Estimated); Status verified 2016-12

CONDITIONS: Urinary Bladder Neurogenic Dysfunction
Keywords: neurogenic detrusor overactivity; detrusor sphincter dyssynergia; compliance; video urodynamic; spinal cord injury
MeSH Terms: conditions — Urinary Bladder, Neurogenic; Patient Compliance; Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- patients with SCI for at least 5 years: Ages Eligibility: minimum 18 years Genders Eligibility: female and male
  Interventions: Other: Video-urodynamic examination

INTERVENTIONS:
Other: Video-urodynamic examination

SUMMARY:
Most patients with spinal cord injury suffer from bladder dysfunction which may - especially in the long-term - impair renal function. Improved treatment during the last decades improved life expectancy and quality of life. This study evaluates the bladder function in the long-term after spinal cord injury.

DETAILED DESCRIPTION:
Bladder dysfunction is a common consequence of spinal cord injury and depends on the completeness and the level of the lesion. Patients with suprasacral injury usually suffer from neurogenic detrusor overactivity mostly combined with detrusor sphincter dyssynergia. Without adequate treatment, this adverse combination puts the upper urinary tract at risk due to high intravesical pressure often causing vesico-ureteral reflux. Based on improved therapeutic options in the last decades, life expectancy and quality of life constantly increased in spinal cord injury patients. The investigators aim to evaluate the bladder function in the long-term after spinal cord injury.

ELIGIBILITY:
Inclusion Criteria:

* Spinal cord injury for at least 5 years
* Neurogenic lower urinary tract dysfunction
* Written informed consent

Exclusion Criteria:

* Lower urinary tract dysfunction due to other causes than spinal cord injury

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Ages Eligibility: minimum 18 years old Genders Eligibility: female and male
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2010-01; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Urodynamic evaluation | 5 years after SCI, yearly thereafter (participants are followed until death)
  Max. cystometric capacity, compliance, detrusor leak point pressure

SECONDARY OUTCOMES:
secondary complications | 5 years after SCI, yearly thereafter (participants are followed until death)
  recurrent tract infection, deterioration of the upper urinary tract
imaging of the upper urinary tract | 5 years after SCI, yearly thereafter (participants are followed until death)
  videocystography, ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Jens Wöllner, Dr. med., Principal Investigator — Balgrist University Hospital
Locations (1):
- Spinal Cord Injury Center & Research, University of Zürich, Balgrist University Hospital, Zurich, Canton of Zurich, Switzerland